CLINICAL TRIAL: NCT04969991
Title: A Phase 2, Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Efficacy of Varespladib in Patients Hospitalized With Severe COVID 19 Caused by SARS-CoV-2
Brief Title: Study of Varespladib in Patients Hospitalized With Severe COVID-19
Acronym: STAIRS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Part 2 of the study was paused on 03-May-2022 due to slow enrollment following low infection rates and hospitalizations of patients with severe COVID-19, and did not recommence prior to study closure (early termination) on 22-Nov-2022.
Sponsor: Ophirex, Inc. (Industry)
Collaborators: Premier Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OPX-PR-02; W81XWH20C0066 (Other: USA Medical Research Acquisition Activity)
Record Dates: First submitted 2021-07-08; First posted 2021-07-21 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-04

CONDITIONS: Coronavirus Disease 2019; Disease Caused by Severe Acute Respiratory Syndrome Coronavirus 2
Keywords: acute respiratory distress syndrome; varespladib; LY333013; severe acute respiratory syndrome coronavirus 2; coronavirus disease 2019; ARDS
MeSH Terms: conditions — COVID-19; Respiratory Distress Syndrome | interventions — varespladib; varespladib methyl

STUDY DESIGN:
Intervention Model Description: The study will be conducted in 2 parts. Both parts will be randomized and double-blind. Part 1 will be dose-finding in 4 parallel treatment groups randomized to treatment with varespladib (at 250 mg once daily [QD], twice daily [BID], or three times daily [TID] [total doses of 250, 500, or 750 mg/day]) or placebo in a 5:5:5:3 ratio. After all participants in Part 1 have completed Day 28, a data safety monitoring board (DSMB) will review the safety results from Part 1 and will recommend the dose regimen to be used in Part 2. Part 2 will randomize an additional 72 participants to the dose regimen selected from Part 1 or placebo in a 1:1 ratio.
  In both parts of the study, eligible participants will be enrolled and randomized to receive either varespladib or placebo in addition to institutional standard of care for 7 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All participants, investigators, and study personnel involved in the conduct of the study, including data management, will be blinded to treatment assignment with the exception of a specified unblinded statistician, an unblinded pharmacist at each clinical site, a programmer from the contract research organization (CRO) who will have access to the randomization code, and the DSMB.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Varespladib: 250 mg QD + Placebo + placebo (Experimental): For 7 days, and in addition to institutional standard of care, participants will take 250 mg varespladib in the morning. In order to maintain the blind, they will also take 1 placebo tablet in the afternoon and 1 placebo tablet in the evening.
  Interventions: Drug: Varespladib; Drug: Placebo
- Varespladib: 250 mg BID + placebo (Experimental): For 7 days, and in addition to institutional standard of care, participants will take 250 mg varespladib in the morning and in the evening. In order to maintain the blind, they will also take 1 placebo tablet in the afternoon.
  Interventions: Drug: Varespladib; Drug: Placebo
- Varespladib: 250 mg TID (Experimental): For 7 days, and in addition to institutional standard of care, participants will take 250 mg varespladib in the morning, in the afternoon, and in the evening.
  Interventions: Drug: Varespladib
- Placebo (Placebo Comparator): For 7 days, and in addition to institutional standard of care, participants will take 1 placebo tablet in the morning, in the afternoon, and in the evening.
  Interventions: Drug: Placebo
- Varespladib: 250mg BID (Part 2 of trial) (Experimental): Dose chosen for Part 2 was twice a day dosing. For 7 days, and in addition to institutional standard of care, participants will take 250 mg varespladib in the morning, and in the evening.
  Interventions: Drug: Varespladib
- Placebo (Part 2 of trial) (Placebo Comparator): For 7 days, and in addition to institutional standard of care, participants will take 1 placebo tablet in the morning, and in the afternoon.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varespladib — 250 mg immediate-release oblong, white, film-coated tablet for oral administration
  Other Names: LY333013
  Arms: Varespladib: 250 mg BID + placebo; Varespladib: 250 mg QD + Placebo + placebo; Varespladib: 250 mg TID; Varespladib: 250mg BID (Part 2 of trial)
Drug: Placebo — Oral formulation matched to the oral varespladib tablet
  Arms: Placebo; Placebo (Part 2 of trial); Varespladib: 250 mg BID + placebo; Varespladib: 250 mg QD + Placebo + placebo

SUMMARY:
This is a 2-part, multi-center, randomized, double-blind, placebo-controlled, phase 2 study designed to evaluate the safety, tolerability, and efficacy of oral varespladib, in addition to standard of care, in patients hospitalized with severe COVID-19 caused by SARS-CoV-2.

DETAILED DESCRIPTION:
The goals of this 2-part, multi-center, randomized, double-blind, placebo-controlled, phase 2 study are to define a safe dose for the population and to assess the safety, tolerability, and efficacy of orally dosed varespladib to improve survival without respiratory failure in patients hospitalized with severe coronavirus disease 2019 (COVID-19), when given in addition to the institutional standard of care therapy.

Mortality rates of COVID-19 are strongly linked to acute respiratory distress syndrome (ARDS) which may be, additionally, correlated with elevations of secretory phospholipase 2 (sPLA2) and widespread loss of functioning lung tissue. Upregulation of sPLA2 is thought to be involved in the dysregulated inflammatory cascade pathways (increased markers of immune activation, also known as cytokine release syndrome) and enzymatic degradation of lung surfactant linked to the development of ARDS. It is believed that treatment with varespladib, a potent inhibitor of sPLA2, might prevent or mitigate progression of pulmonary dysfunction in COVID-19 patients by two mechanisms: suppression of sPLA2-induced inflammation and, uniquely, preservation of pulmonary surfactant by direct inhibition of the enzyme responsible for surfactant phospholipid degradation: sPLA2.

Data from previous phase 2 clinical trials of varespladib suggested it had potential to reduce mortality in severely septic patients with ARDS, particularly when treatment was initiated within 18 hours of identification of organ failure.

The study will be conducted in two parts. Both parts will be randomized and double-blind. Part 1 will be dose-finding in four parallel treatment groups randomized to treatment with varespladib (at 250 mg once daily [QD], twice daily [BID], or three times daily [TID] [250, 500, or 750 mg/day]) or placebo in a 5:5:5:3 ratio. After all participants in Part 1 have completed Day 28, a data safety monitoring board (DSMB) will review the safety results from Part 1, including all available safety data through Day 60, and will recommend the dose regimen to be used in Part 2. Part 2 will randomize an additional 72 participants to the dose regimen selected from Part 1 or placebo in a 1:1 ratio.

In both parts of the study, eligible participants will be enrolled and randomized to receive active varespladib or placebo in addition to institutional standard of care for 7 days.

Participants will be assessed daily per standard of care while hospitalized and on a regular basis after discharge. The Day 1, 4, 7, 14, and 28 visits will be performed in person (either at the hospital/site or via a home health provider) to assess safety, obtain blood and urine samples for laboratory tests, and obtain clinical outcome data. The Day 2, 3, 5, 6, 8, 9, 10, 11, 12, 13, 15, 16, 17, 18, 19, 20, 21, 45, and 60 visits for discharged participants may be conducted by phone or via electronic patient-reported outcome (ePRO) devices.

Efficacy will be assessed by respiratory failure-free survival at Day 28. Safety will be assessed by evaluating adverse events (AEs), vital sign measurements, use of oxygen therapies, changes in levels of biomarkers, clinical laboratory test results, electrocardiograms (ECGs), physical examination findings, and concomitant medications and therapies. A DSMB will evaluate safety data at specified intervals during both parts of the trial.

Pharmacokinetic (PK) samples will be drawn from all participants in Part 1 and in a subset of approximately 14 participants in Part 2 in order to enable estimation of PK parameters in approximately 22 participants receiving active treatment with varespladib.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is hospitalized with severe COVID-19 illness, defined in accordance with the Food and Drug Administration (FDA) Guidance for Industry - COVID-19: Developing Drugs and Biological Products for Treatment or Prevention (May 2020):

   a. Severe illness:

   i. Symptoms suggestive of severe systemic illness with COVID-19, which could include any symptom of moderate illness or shortness of breath at rest, or respiratory distress

   ii. Clinical signs indicative of severe systemic illness with COVID-19, such as respiratory rate ≥30 per minute, heart rate ≥125 per minute, SpO₂ ≤93% on room air at sea level or partial pressure of oxygen PaO₂/fraction of inspired oxygen FiO₂ <300.
2. Participant has a positive virologic nucleic acid amplification test (NAAT) indicating SARS-CoV-2 infection in a sample collected <72 hours prior to randomization.
3. Participant is between the ages of 18 and 80 years at the time of enrollment.
4. Participant provides informed consent prior to initiation of any study procedures.
5. Participant agrees to not participate in another clinical trial for the treatment of COVID 19 or SARS-CoV-2 through Day 28.
6. Participant has adequate hematologic status (in the absence of transfusion and growth factor support for at least 28 days), defined as follows:

   1. Absolute neutrophil count (ANC) ≥1.5 × 10⁹/L
   2. Platelet count ≥75 × 10⁹/L
   3. Hemoglobin ≥9 g/dL.
7. Participant has an Eastern Cooperative Oncology Group (ECOG) performance score of 0-2.

Exclusion Criteria:

1. Participant has mild, moderate, or critical COVID-19 defined in accordance with the FDA Guidance for Industry:

   a. Mild COVID-19:

   i. Symptoms of mild illness with COVID-19 that could include fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms, without shortness of breath or dyspnea

   ii. No clinical signs indicative of moderate, severe, or critical severity

   b. Moderate COVID-19:

   i. Symptoms of moderate illness with COVID-19, which could include any symptom of mild illness (fever, cough, sore throat, malaise, headache, muscle pain, gastrointestinal symptoms) or shortness of breath with exertion

   ii. Clinical signs suggestive of moderate illness with COVID-19, such as respiratory rate ≥20 breaths per minute, peripheral oxygen saturation (SpO₂) >93% on room air at sea level, heart rate ≥90 beats per minute

   iii. No clinical signs indicative of severe or critical illness

   c. Critical COVID-19:

   i. Respiratory failure defined based on resource utilization requiring at least one of the following:
   * Endotracheal intubation and mechanical ventilation
   * Oxygen delivered by high-flow nasal cannula ([HFNC] heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥0.5)
   * Noninvasive positive pressure ventilation
   * ECMO, or
   * Clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting of resource limitation)

   ii. Shock (defined by systolic blood pressure <90 mmHg, or diastolic blood pressure <60 mmHg or requiring vasopressors)

   iii. Multi-organ dysfunction/failure.
2. Participant has taken investigational medications within 7 days or 5 half-lives prior to enrollment, whichever is shorter.
3. Participant has required any new form of sedation, anxiolysis or central nervous system (CNS) depressant within the 48 hours prior to enrollment that would interfere with neurologic assessments at enrollment.
4. Has history of cerebrovascular accident or intracranial bleeding of any kind, acute coronary syndrome, myocardial infarction, or severe pulmonary hypertension.
5. Participant has chronic respiratory failure not associated with COVID-19, defined as prior need for home oxygen, need for home noninvasive positive-pressure ventilation (NIPPV) for reasons other than isolated sleep apnea, or other signs of chronic respiratory failure, in the investigator's judgment.
6. Upper gastrointestinal (GI) bleed evidenced by hematemesis, "coffee-ground" emesis or nasogastric aspirate, or hematochezia thought to originate from upper GI tract.
7. Participant has abnormal liver function defined as any 2 of the following at screening:

   1. Total bilirubin ≥2 × ULN
   2. Alanine aminotransferase (ALT) ≥3 × ULN
   3. Aspartate aminotransferase (AST) ≥3 × ULN
   4. Alkaline phosphatase (ALP) >3 × ULN
   5. Gamma-glutamyl transferase (GGT) >3 × ULN
8. Participant has an estimated glomerular filtration rate (eGFR) <60 mL/min.
9. Participant has a known allergy or significant adverse reaction to varespladib-methyl or related compounds.
10. Participant is considered by the investigator to be unable to comply with protocol requirements due to geographic considerations, psychiatric disorders, or other compliance concerns; or has any serious medical condition or clinically significant laboratory, ECG, vital sign, or physical examination abnormality that would prevent study participation or place the participant at significant risk, as judged by the Investigator.
11. Participant is breast-feeding, pregnant, has a positive serum hCG pregnancy test, or is not willing to use a highly effective method of contraception for 14 days after treatment. Highly effective methods of contraception are as follows:

    1. Combined (estrogen- and progestogen-containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, or transdermal)
    2. Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, or implantable)
    3. Intrauterine device, intrauterine hormone-releasing system
    4. Bilateral tubal occlusion
    5. Vasectomized partner
    6. Sexual abstinence
    7. Double-barrier method (condoms, sponge, diaphragm, with spermicidal jellies, or cream).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2022-02-11 (Actual); Study Completion 2022-11-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Ventura Clinical Trials, Ventura, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Westchester Research Center at Westchester General Hospital, Miami, Florida
  - Franciscan Alliance, Munster, Indiana
  - The Brigham and Women's Hospital Emergency Medicine, Boston, Massachusetts
  - Cooper University Hospital, Camden, New Jersey
  - Ascension St. John Clinical Research Institute, Tulsa, Oklahoma

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rezoagli E, Fumagalli R, Bellani G. Definition and epidemiology of acute respiratory distress syndrome. Ann Transl Med. 2017 Jul;5(14):282. doi: 10.21037/atm.2017.06.62. PMID 28828357
- [Background] Englert JA, Bobba C, Baron RM. Integrating molecular pathogenesis and clinical translation in sepsis-induced acute respiratory distress syndrome. JCI Insight. 2019 Jan 24;4(2):e124061. doi: 10.1172/jci.insight.124061. PMID 30674720
- [Background] Mirastschijski U, Dembinski R, Maedler K. Lung Surfactant for Pulmonary Barrier Restoration in Patients With COVID-19 Pneumonia. Front Med (Lausanne). 2020 May 22;7:254. doi: 10.3389/fmed.2020.00254. eCollection 2020. No abstract available. PMID 32574339
- [Background] Griffiths MJD, McAuley DF, Perkins GD, Barrett N, Blackwood B, Boyle A, Chee N, Connolly B, Dark P, Finney S, Salam A, Silversides J, Tarmey N, Wise MP, Baudouin SV. Guidelines on the management of acute respiratory distress syndrome. BMJ Open Respir Res. 2019 May 24;6(1):e000420. doi: 10.1136/bmjresp-2019-000420. eCollection 2019. PMID 31258917
- [Background] Huang C, Wang Y, Li X, Ren L, Zhao J, Hu Y, Zhang L, Fan G, Xu J, Gu X, Cheng Z, Yu T, Xia J, Wei Y, Wu W, Xie X, Yin W, Li H, Liu M, Xiao Y, Gao H, Guo L, Xie J, Wang G, Jiang R, Gao Z, Jin Q, Wang J, Cao B. Clinical features of patients infected with 2019 novel coronavirus in Wuhan, China. Lancet. 2020 Feb 15;395(10223):497-506. doi: 10.1016/S0140-6736(20)30183-5. Epub 2020 Jan 24. PMID 31986264
- [Background] Wang D, Hu B, Hu C, Zhu F, Liu X, Zhang J, Wang B, Xiang H, Cheng Z, Xiong Y, Zhao Y, Li Y, Wang X, Peng Z. Clinical Characteristics of 138 Hospitalized Patients With 2019 Novel Coronavirus-Infected Pneumonia in Wuhan, China. JAMA. 2020 Mar 17;323(11):1061-1069. doi: 10.1001/jama.2020.1585. PMID 32031570
- [Background] Yang X, Yu Y, Xu J, Shu H, Xia J, Liu H, Wu Y, Zhang L, Yu Z, Fang M, Yu T, Wang Y, Pan S, Zou X, Yuan S, Shang Y. Clinical course and outcomes of critically ill patients with SARS-CoV-2 pneumonia in Wuhan, China: a single-centered, retrospective, observational study. Lancet Respir Med. 2020 May;8(5):475-481. doi: 10.1016/S2213-2600(20)30079-5. Epub 2020 Feb 24. PMID 32105632
- [Background] Gandhi RT, Lynch JB, Del Rio C. Mild or Moderate Covid-19. N Engl J Med. 2020 Oct 29;383(18):1757-1766. doi: 10.1056/NEJMcp2009249. Epub 2020 Apr 24. No abstract available. PMID 32329974
- [Background] Abraham E, Naum C, Bandi V, Gervich D, Lowry SF, Wunderink R, Schein RM, Macias W, Skerjanec S, Dmitrienko A, Farid N, Forgue ST, Jiang F. Efficacy and safety of LY315920Na/S-5920, a selective inhibitor of 14-kDa group IIA secretory phospholipase A2, in patients with suspected sepsis and organ failure. Crit Care Med. 2003 Mar;31(3):718-28. doi: 10.1097/01.CCM.0000053648.42884.89. PMID 12626975
- [Background] Ware J Jr, Kosinski M, Keller SD. A 12-Item Short-Form Health Survey: construction of scales and preliminary tests of reliability and validity. Med Care. 1996 Mar;34(3):220-33. doi: 10.1097/00005650-199603000-00003. PMID 8628042
- [Background] Food and Drug Administration. Guidance for Industry on COVID-19: Developing Drugs and Biological Products for Treatment or Prevention, May 2020.
- See also: COVID-19 Clinical management: living guidance — https://www.who.int/publications/i/item/WHO-2019-nCoV-clinical-2021-2
- See also: In patients of COVID-19, what are the symptoms and clinical features of mild and moderate cases? — https://www.cebm.net/covid-19/in-patients-of-covid-19-what-are-the-symptoms-and-clinical-features-of-mild-and-moderate-case/

RESULTS

PARTICIPANT FLOW:
Period: Part 1
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Started | 5 | 5 | 5 | 3
Completed | 4 | 4 | 5 | 3
Not Completed | 1 | 1 | 0 | 0
Period: Part 2
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Started | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 1
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo | Total
Number analyzed (Participants) | 5 | 5 | 5 | 3 | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.0 (22.9) | 42.6 (17.1) | 48.6 (8.9) | 62.0 (15.7) | 50.4 (17.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 2 | 1 | 9
  Male | 1 | 3 | 3 | 2 | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 3 | 3 | 2 | 12
  Not Hispanic or Latino | 1 | 2 | 2 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1 | 2
  White | 5 | 3 | 5 | 2 | 15
  More than one race | 0 | 1 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants Alive and Free of Respiratory Failure at Day 28
Description: The proportion of respiratory failure-free surviving participants in each Part 2 treatment group at Day 28 will be analyzed using the Mantel-Haenszel stratum-weighted estimator with treatment as a factor. Respiratory failure is defined based on resource utilization requiring at least one of the following:
  * Endotracheal intubation and mechanical ventilation
  * Oxygen delivered by high-flow nasal cannula ([HFNC] heated, humidified, oxygen delivered via reinforced nasal cannula at flow rates >20 L/min with fraction of delivered oxygen ≥0.5)
  * Noninvasive positive pressure ventilation
  * ECMO, or
  * Clinical diagnosis of respiratory failure (i.e., clinical need for one of the preceding therapies, but preceding therapies not able to be administered in setting because of resource limitation)
Time Frame: Baseline to Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 4 | 4 | 3 | 3

2. Secondary Outcome: Proportion of Subjects Using HFNC Within the First 28 Days After Randomization
Description: The proportion of subjects using HFNC within the first 28 days after randomization.
Time Frame: From randomization through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 1 | 2 | 0

3. Secondary Outcome: Proportion of Subjects Using Noninvasive Respiratory Support Within the First 28 Days After Randomization
Description: Proportion of subjects using noninvasive respiratory support within the first 28 days after randomization.
Time Frame: From randomization through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 1 | 1 | 0 | 0

4. Secondary Outcome: Proportion of Subjects Using Mechanical Ventilation Within the First 28 Days After Randomization
Description: Proportion of subjects using mechanical ventilation within the first 28 days after randomization.
Time Frame: From randomization through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 1 | 0 | 1 | 0

5. Secondary Outcome: Number of Days of Oxygen Support Through Day 28 After Randomization
Description: Number of days of oxygen support through Day 28 after randomization.
Time Frame: From randomization through Day 28
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
days | 9 (11) | 6 (8) | 12 (11) | 11 (15)

6. Secondary Outcome: Proportion of Participants Remaining Free of Mechanical Ventilation or ECMO Throughout the 28 Days After Randomization
Description: Proportion of participants remaining free of mechanical ventilation or ECMO throughout the 28 days after randomization.
Time Frame: From randomization through Day 28
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 4 | 5 | 4 | 3

7. Secondary Outcome: Proportion of Subjects With All-cause Mortality Through Day 60
Description: Proportion of subjects who experience all-cause mortality from randomization through Day 60.
Time Frame: From randomization through Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 1 | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Change in Body Temperature
Description: Number of participants with change in body temperature from providing informed consent through Day 60.
Time Frame: From providing informed consent through Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
Number analyzed (Participants) | 5 | 5 | 5 | 3
Participants | 0 | 0 | 1 | 0

9. Other Pre Specified Outcome: Participant-reported Quality-of-life Assessment Using the 12-item Short Form Survey (SF-12) at Day 28 After Randomization
Description: Changes from baseline to Day 28 in SF-12 scores, which range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Time Frame: Day 28
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Activity of sPLA2 Within Blood Samples Collected as Clinically Required From Treatment Initiation to Day 28 After Randomization
Description: Changes in observed sPLA2 values
Time Frame: From treatment initiation through Day 28
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Changes in PK Parameters: Area-under-the-curve (AUC)
Description: Change in AUC from Day 1 through Day 3
Time Frame: Day 1 through Day 3
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Changes in PK Parameters: Maximum Concentration (Cmax)
Description: Change in Cmax from Day 1 through Day 3
Time Frame: Day 1 through Day 3
Reporting Status: Not Posted

13. Other Pre Specified Outcome: Changes in PK Parameters: Time of Cmax (Tmax)
Description: Change in Tmax from Day 1 through Day 3
Time Frame: Day 1 through Day 3
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Treatment-emergent AEs were events that occurred or worsened on or after the first dose of study intervention and prior to the 30 days after last administration of study intervention. AEs were reported through 60 days after randomization.
Arm/Group | Varespladib: 250 mg QD + Placebo + Placebo | Varespladib: 250 mg BID + Placebo | Varespladib: 250 mg TID | Placebo
All-Cause Mortality (participants affected / at risk) | 1/5 | 0/5 | 0/5 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/5 | 1/5 | 0/5 | 0/3
Other Adverse Events (participants affected / at risk) | 0/5 | 2/5 | 0/5 | 0/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varespladib: 250 mg QD + Placebo + Placebo (N=5) | Varespladib: 250 mg BID + Placebo (N=5) | Varespladib: 250 mg TID (N=5) | Placebo (N=3)
Progression of COVID 19 (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism & COVID 19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Varespladib: 250 mg QD + Placebo + Placebo (N=5) | Varespladib: 250 mg BID + Placebo (N=5) | Varespladib: 250 mg TID (N=5) | Placebo (N=3)
Hypotension (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transaminases Increased (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-02-28): https://cdn.clinicaltrials.gov/large-docs/91/NCT04969991/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/91/NCT04969991/SAP_001.pdf